CLINICAL TRIAL: NCT00357084
Title: A Phase II Study to Evaluate Efficacy and Tolerability of Methotrexate in Combination With Glucocorticoids for the Treatment of Newly Diagnosed Acute Graft-Versus-Host Disease After Nonmyeloablative Hematopoietic Cell Transplantation
Brief Title: Methotrexate and Glucocorticoids in Treating Patients With Newly Diagnosed Acute Graft-Versus-Host Disease After Donor Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Marco B. Mielcarek, Fred Hutchinson Cancer Research Center
Purpose: Supportive Care
Other Study IDs: 1978.00; FHCRC-1978.00; CDR0000488486 (Registry Identifier: PDQ)
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Cancer
Keywords: graft versus host disease; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; atypical chronic myeloid leukemia; blastic phase chronic myelogenous leukemia; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia; chronic eosinophilic leukemia; chronic idiopathic myelofibrosis; chronic myelomonocytic leukemia; chronic neutrophilic leukemia; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; disseminated neuroblastoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; juvenile myelomonocytic leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; nodal marginal zone B-cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; poor prognosis metastatic gestational trophoblastic tumor; previously treated childhood rhabdomyosarcoma; previously treated myelodysplastic syndromes; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult Burkitt lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent/refractory childhood Hodgkin lymphoma; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood rhabdomyosarcoma; recurrent childhood small noncleaved cell lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent small lymphocytic lymphoma; recurrent Wilms tumor and other childhood kidney tumors; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; refractory multiple myeloma; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; splenic marginal zone lymphoma; stage I multiple myeloma; stage II multiple myeloma; stage II ovarian epithelial cancer; stage III adult Burkitt lymphoma; stage III adult Hodgkin lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III multiple myeloma; stage III small lymphocytic lymphoma; stage III malignant testicular germ cell tumor; stage IV adult Burkitt lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV chronic lymphocytic leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; Waldenstrom macroglobulinemia; childhood myelodysplastic syndromes
MeSH Terms: conditions — Neoplasms; Graft vs Host Disease; Congenital Abnormalities; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelomonocytic, Juvenile; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Recurrence; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Wilms Tumor; Leukemia, Hairy Cell; Multiple Myeloma; Carcinoma, Ovarian Epithelial; Testicular Neoplasms; Waldenstrom Macroglobulinemia | interventions — Methotrexate; Methylprednisolone; Prednisone

INTERVENTIONS:
Drug: methotrexate
Drug: methylprednisolone
Drug: prednisone

SUMMARY:
RATIONALE: Methotrexate and glucocorticoid therapy, such as prednisone or methylprednisolone, may be an effective treatment for acute graft-versus-host disease caused by a donor stem cell transplant.

PURPOSE: This phase II trial is studying how well giving methotrexate together with glucocorticoids works in treating patients with newly diagnosed acute graft-versus-host disease after donor stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine, within the limits of a phase II study, whether low-dose methotrexate can accelerate withdrawal of glucocorticoids and decrease nonrelapsing mortality in patients with newly diagnosed acute graft-versus-host disease (GVHD) who have undergone nonmyeloablative allogeneic hematopoietic stem cell transplantation (HSCT).
* Determine the tolerability of low-dose methotrexate and glucocorticoids in treating newly diagnosed acute GVHD in these patients.

OUTLINE: This is a cohort study. Patients receive concurrent low-dose methotrexate and a glucocorticoid for treatment of acute graft-versus-host disease (GVHD).

Patients receive the first dose of methotrexate IV ≥ 12 hours before initiation of glucocorticoid treatment (if glucocorticoid treatment has not been initiated) and the second dose 72 hours after dose 1. Patients then receive subsequent doses of methotrexate IV or orally once weekly for up to 1 year* until resolution of GVHD in the absence of recurrent malignancy, refractory or chronic GVHD, administration of secondary treatment for GVHD, or unacceptable toxicity.

NOTE: *Treatment with low-dose MTX may continue beyond 1 year at the discretion of the managing physician.

Patients receive glucocorticoid therapy comprising prednisone or methylprednisolone IV twice daily until objective evidence of improvement in GVHD manifestation. Patients with resolved or significantly improved GVHD receive treatment for 10 days followed by an accelerated taper for a total of 72 days of treatment in case of no flare up of GVHD during the glucocorticoid taper. Patients with exacerbation or recurrence of GVHD during the accelerated taper are treated for ≥ 1 week before resuming a less rapid taper. Patients who develop GVHD progression or primary refractory GVHD may receive secondary systemic therapy at the discretion of the managing physician.

After completion of study treatment, patients are followed at 1 year and then annually thereafter.

PROJECTED ACCRUAL: A total of 53 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed acute graft-versus-host disease (GVHD)
* Has undergone nonmyeloablative allogeneic hematopoietic stem cell transplantation (HSCT) from an HLA-matched related or unrelated donor ≥ 14 days ago
* Treatment of GVHD with glucocorticoids indicated by 1 of the following criteria:

  * Initial treatment with prednisone or methylprednisolone at 2 mg/kg indicated (in the judgement of attending physician) by any of the following:

    * Severity of GVHD requires hospitalization
    * GVHD manifestations include symptoms other than anorexia, nausea, and vomiting
    * GVHD begins within 2-3 weeks after HSCT
    * GVHD manifestations progress rapidly from 1 day to the next before treatment
  * Initial treatment with prednisone or methylprednisolone at 1 mg/kg did not produce adequate clinical improvement within the first 4 days (in the judgement of attending physician)
* No pleural effusion or ascites (i.e., free-flowing fluid by lateral decubitus views)

  * Mere blunting of costo-phrenic angles on a posterior anterior chest x-ray is not sufficient
* No GVHD after donor lymphocyte infusion
* No hallmarks of chronic GVHD
* No bronchiolitis obliterans

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of study treatment
* No severe mucositis (grade 3 or 4) indicated by erythema, edema, or ulcerations requiring hydration, parenteral nutritional support, or intubation or resulting in aspiration pneumonia
* Absolute neutrophil count ≥ 1,500/mm^3
* Bilirubin ≤ 2 times upper limit of normal (ULN) (unless abnormality attributable to GVHD)
* AST and ALT ≤ 2 times ULN (unless abnormality attributable to GVHD)
* Creatinine clearance ≥ 50 mL/min

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior prednisone or methylprednisolone at 2 mg/kg for > 72 hours or at 1 mg/kg for > 96 hours
* Concurrent topical therapy, including psoralen and ultraviolet A irradiation (PUVA), glucocorticoid creams, oral beclomethasone dipropionate, topical azathioprine, or ophthalmic glucocorticoids allowed
* No other concurrent treatment for GVHD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2006-05; Primary Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients treated with a methylprednisolone-equivalent glucocorticoid dose ≤ 0.75 mg/kg on day 28 after initiation of systemic glucocorticoid therapy for acute graft-versus-host disease (GVHD)

SECONDARY OUTCOMES:
Proportion of patients in whom methotrexate (MTX) had to be discontinued because of toxicity
Incidence of severe acute GVHD (grades III or IV)
Incidence of extensive chronic GVHD
Incidence of secondary systemic immunosuppressive therapy
Cumulative corticosteroid use over 1 year
Nonrelapsing mortality at 1 year
Incidence of invasive mold infections
Incidence of recurrent/progressive malignancy
Cumulative dose of methylprednisolone-equivalent treatment during the first 8 weeks after enrollment in patients who survive to day 56

CONTACTS AND LOCATIONS:
Overall Officials: Marco B. Mielcarek, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States